CLINICAL TRIAL: NCT04039503
Title: Randomized, Phase 3, Double-blind Trial Comparing the Effect of the Addition of Tirzepatide Versus Placebo in Patients With Type 2 Diabetes Inadequately Controlled on Insulin Glargine With or Without Metformin
Brief Title: A Study of Tirzepatide (LY3298176) Versus Placebo in Participants With Type 2 Diabetes Inadequately Controlled on Insulin Glargine With or Without Metformin
Acronym: SURPASS-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16998; I8F-MC-GPGI (Other: Eli Lilly and Company); 2019-000860-99 (EudraCT Number)
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12-01

CONDITIONS: Type 2 Diabetes
Keywords: glucose-dependent insulinotropic polypeptide (GIP); glucagon-like peptide-1 (GLP-1); GIP/GLP-1 dual receptor agonist; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Tirzepatide (Experimental): 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Placebo administered SC once a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC as add-on to the pre-trial background medication.
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Placebo — Administered SC as add-on to the pre-trial background medication.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and efficacy of the study drug tirzepatide to placebo in participants with type 2 diabetes that are already on insulin glargine, with or without metformin. Participants will administer tirzepatide or placebo along with their previous glucose lowering medications. The study will last approximately 47 weeks and may include about 23 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus (T2DM) and have been treated with insulin glargine (U100), once daily with or without metformin ≥3 months prior to screening visit.
* Have HbA1c between ≥7.0% and ≤10.5%.
* Have a stable weight (± 5%) for at least 3 months before screening.
* Have a body mass index (BMI) ≥23 kilograms per meter squared (kg/m²) at screening.

Exclusion Criteria:

* Have type 1 diabetes mellitus.
* Have had chronic or acute pancreatitis any time prior to study entry.
* Have proliferative diabetic retinopathy or diabetic maculopathy or nonproliferative diabetic retinopathy requiring acute treatment.
* Have disorders associated with slowed emptying of the stomach, or have had any stomach surgeries for the purpose of weight loss.
* Have an estimated glomerular filtration rate <30 mL/minute/1.73 m² [for participants on metformin, estimated glomerular filtration rate <45 mL/min/1.73 m2 (or lower than the country-specific threshold for using the protocol-required dose of metformin per local label)]
* Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months.
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2.
* Have been taking weight loss drugs, including over-the-counter medications during the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (48):
- United States (5):
  - Valley Endocrine, Fresno, Fresno, California
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Manhattan Medical Research, New York, New York
  - Intend Research, Norman, Oklahoma
- Czechia (7):
  - Milan Kvapil s.r.o., Příbram, Central Bohemia
  - Diacentrum Brandys n.L. s.r.o., Brandys Nad Labem-Stara Bolesl
  - Diabetologicka ordinace pro dospele, Krnov
  - Diahelp s.r.o., Interni a diabetologicka ambulance, Pardubice
  - Lekarna Dr. Max, Prague
  - Milan Kvapil s.r.o., Prague
  - RESTRIAL s.r.o., Prague
- Germany (10):
  - Praxis Dr. Jörg Lüdemann, Falkensee, Brandenburg
  - Arztpraxis Dr. Cornelia Marck, Pohlheim, Hesse
  - InnoDiab Forschung GmbH, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung Münster GmbH, Münster, North Rhine-Westphalia
  - Praxis Dr. Kempe - Dr. Stemler, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Schwerpunktpraxis Diabetes, Saint Ingbert-Oberwürzbach, Saarland
  - SMO.MD GmbH, Magdeburg, Saxony-Anhalt
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabetologische Schwerpunktpraxis B. Scholz/Dr. B. Paschen, Hamburg
  - Gemeinschaftspraxis für innere Medizin und Diabetologie, Hamburg
- Japan (10):
  - Kashiwa hospital, Kashiwa, Chiba
  - Manda Hospital, Sapporo, Hokkaido
  - Takai Naika Clinic, Kamakura, Kanagawa
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Tokyo Center Clinic, Chuo-ku, Tokyo
  - Tokyo Clinical Trial Centre Fukuwa Clinic, Chuo-ku, Tokyo
  - The Institute for Adult Diseases, Asahi Life Foundation, Chuou-ku, Tokyo
  - Sato Naika Clinic, Ōta-ku, Tokyo
  - Jinnouchi Hospital, Kumamoto
- Poland (4):
  - Centrum Medyczne AMED, Warsaw, Masovian Voivodeship
  - NZOZ ZDROWIE Osteo-Medic, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych, PI House, Gdansk, Pomeranian Voivodeship
  - NZOZ Przychodnia Specjalistyczna MEDICA, Lublin
- Puerto Rico (2):
  - Centro de Endocrinologia y Nutricion del Turabo, Caguas, PR
  - Manati Center for Clinical Research Inc, Manatí, PR
- Slovakia (5):
  - Ambulancia vnútorného lekárstva Hnúša (Diabetes care), Hnúšťa
  - Sin Azucar, Malacky
  - Dia-Clarus.s.r.o., Prievidza
  - JAL, Trnava
  - Medivasa, s.r.o., Žilina
- Spain (5):
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital de la Ribera, Alzira, Valencia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Infanta Luisa, Seville
  - Hospital Universitari i Politecnic La Fe-ENDO, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] De Block C, Peleshok J, Wilding JPH, Kwan AYM, Rasouli N, Maldonado JM, Wysham C, Liu M, Aleppo G, Benneyworth BD. Post Hoc Analysis of SURPASS-1 to -5: Efficacy and Safety of Tirzepatide in Adults with Type 2 Diabetes are Independent of Baseline Characteristics. Diabetes Ther. 2025 Jan;16(1):43-71. doi: 10.1007/s13300-024-01660-0. Epub 2024 Nov 12. PMID 39531161
- [Derived] Boye KS, Sapin H, Dong W, Williamson S, Lee CJ, Thieu VT. Improved Glycaemic and Weight Management Are Associated with Better Quality of Life in People with Type 2 Diabetes Treated with Tirzepatide. Diabetes Ther. 2023 Nov;14(11):1867-1887. doi: 10.1007/s13300-023-01457-7. Epub 2023 Sep 5. PMID 37668888
- [Derived] Boye KS, Thieu VT, Sapin H, Lee CJ, Lando LF, Brown K, Bray R, Wiese RJ, Patel H, Rodriguez A, Yu M. Patient-Reported Outcomes in People with Type 2 Diabetes Receiving Tirzepatide in the SURPASS Clinical Trial Programme. Diabetes Ther. 2023 Nov;14(11):1833-1852. doi: 10.1007/s13300-023-01451-z. Epub 2023 Aug 1. PMID 37526908
- [Derived] Sattar N, McGuire DK, Pavo I, Weerakkody GJ, Nishiyama H, Wiese RJ, Zoungas S. Tirzepatide cardiovascular event risk assessment: a pre-specified meta-analysis. Nat Med. 2022 Mar;28(3):591-598. doi: 10.1038/s41591-022-01707-4. Epub 2022 Feb 24. PMID 35210595
- [Derived] Dahl D, Onishi Y, Norwood P, Huh R, Bray R, Patel H, Rodriguez A. Effect of Subcutaneous Tirzepatide vs Placebo Added to Titrated Insulin Glargine on Glycemic Control in Patients With Type 2 Diabetes: The SURPASS-5 Randomized Clinical Trial. JAMA. 2022 Feb 8;327(6):534-545. doi: 10.1001/jama.2022.0078. PMID 35133415
- See also: A Study of Tirzepatide (LY3298176) Versus Placebo in Participants With Type 2 Diabetes Inadequately Controlled on Insulin Glargine With or Without Metformin — https://trials.lillytrialguide.com/en-US/trial/33Mn9pqfndRwZEPVvpNxDR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Started | 116 | 119 | 120 | 120
Received at Least One Dose of Study Drug | 116 | 119 | 120 | 120
Completed | 109 | 115 | 110 | 117
Not Completed | 7 | 4 | 10 | 3
Not completed — Adverse Event | 3 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 3 | 5 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo | Total
Number analyzed (Participants) | 116 | 119 | 120 | 120 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.50 (9.81) | 60.40 (10.24) | 60.50 (9.92) | 60.00 (9.63) | 60.60 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 47 | 55 | 54 | 211
  Male | 61 | 72 | 65 | 66 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 5 | 5 | 22
  Not Hispanic or Latino | 94 | 95 | 93 | 98 | 380
  Unknown or Not Reported | 18 | 16 | 22 | 17 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 20 | 21 | 22 | 22 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 0 | 6
  White | 95 | 94 | 94 | 97 | 380
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 24 | 24 | 23 | 23 | 94
  Germany | 32 | 32 | 33 | 32 | 129
  Japan | 19 | 21 | 20 | 22 | 82
  Poland | 8 | 9 | 10 | 9 | 36
  Puerto Rico | 2 | 6 | 1 | 3 | 12
  Slovakia | 8 | 7 | 8 | 8 | 31
  Spain | 13 | 15 | 15 | 14 | 57
  United States | 10 | 5 | 10 | 9 | 34
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.30 (0.88) | 8.36 (0.83) | 8.23 (0.86) | 8.37 (0.84) | 8.31 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (10 mg and 15 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Baseline Metformin Use (Yes, No) + Pooled Country + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All randomized participants from who received at least 1 dose study drug and had a baseline and at least 1 post-baseline value, excluding patients discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 113 | 117 | 118
Percentage of HbA1c | -2.59 (0.081) | -2.59 (0.083) | -0.93 (0.079)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.66, 95% CI 2-sided [-1.88 to -1.43]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.65, 95% CI 2-sided [-1.88 to -1.43]

2. Secondary Outcome: Change From Baseline in HbA1c (5 mg)
Description: as for outcome 1
Time Frame: Baseline, Week 40
Population: All randomized participants who received at least one dose of 5 mg tirzepatide, placebo and had a baseline and at least 1 post-baseline value, excluding patients discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Groups:
- 5 mg Tirzepatide: 5 mg tirzepatide administered subcutaneously (SC) once a week.
Arm/Group | 5 mg Tirzepatide | Placebo
Number analyzed (Participants) | 115 | 118
Percentage of HbA1c | -2.23 (0.081) | -0.93 (0.079)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.30, 95% CI 2-sided [-1.52 to -1.07]

3. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Baseline HbA1c Group (<= 8.0%, >8.0%) + Baseline Metformin Use (Yes, No) + Pooled Country + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All randomly assigned participants who took at least 1 dose of study drug and had a baseline and at least 1 post-baseline value, excluding patients discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 115 | 113 | 117 | 118
Kilograms (kg) | -6.2 (0.58) | -8.2 (0.58) | -10.9 (0.59) | 1.7 (0.57)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.8, 95% CI 2-sided [-9.4 to -6.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -9.9, 95% CI 2-sided [-11.5 to -8.3]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -12.6, 95% CI 2-sided [-14.2 to -11.0]

4. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target Value of <7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A.HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 40
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 115 | 113 | 117 | 118
Percentage of Participants | 93.04 | 97.35 | 94.02 | 33.90
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 37.77, 95% CI 2-sided [15.23 to 93.70]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 100.07, 95% CI 2-sided [30.02 to 333.62]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 43.31, 95% CI 2-sided [16.92 to 110.83]

5. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: Fasting serum glucose (FSG) is a test to determine sugar levels in serum sample after an overnight fast. LS Mean was determined by MMRM model with Baseline + Pooled Country + Baseline Metformin Use (Yes, No) + Baseline HbA1c Group (<= 8.0%, >8.0%) + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milligram per Deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 115 | 116 | 118 | 118
milligram per Deciliter (mg/dL) | -61.4 (2.55) | -67.9 (2.55) | -67.7 (2.64) | -38.9 (2.49)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -22.5, 95% CI 2-sided [-29.5 to -15.4]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -29.0, 95% CI 2-sided [-36.0 to -22.0]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -28.8, 95% CI 2-sided [-35.9 to -21.6]

6. Secondary Outcome: Mean Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Postmeal, Midday Premeal, Midday 2-hour Postmeal, Evening Premeal, Evening 2-hour Postmeal and Bedtime. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Baseline HbA1c Group (<= 8.0%, >8.0%) + Baseline Metformin Use (Yes, No) + Pooled Country + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 100 | 99 | 94 | 97
mg/dL | -67.1 (2.05) | -71.7 (2.04) | -73.7 (2.10) | -39.4 (2.07)

7. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss ≥5%
Description: Percentage of Participants who Achieved Weight Loss ≥5%.
Time Frame: Week 40
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 115 | 113 | 117 | 118
Percentage of Participants | 53.91 | 64.60 | 84.62 | 5.93
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 17.15, 95% CI 2-sided [7.55 to 38.93]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 27.24, 95% CI 2-sided [11.87 to 62.55]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 79.61, 95% CI 2-sided [32.76 to 193.44]

8. Secondary Outcome: Percentage Change From Baseline in Daily Mean Insulin Glargine Dose
Description: LS mean was calculated using MMRM model with log (Baseline) + Baseline Metformin Use (Yes, No) + Pooled Country + Baseline HbA1c Group (<= 8.0%, >8.0%) + Treatment + Time + Treatment*Time (Type III sum of squares) as variables.
Time Frame: Baseline, Week 40
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: International Units (IU)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 105 | 103 | 96 | 111
International Units (IU) | 13.0 (7.34) | 8.1 (7.03) | -11.4 (5.85) | 75.0 (11.11)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 10 mg Tirzepatide; Test type: Superiority; Estimate Difference = -35.4, 95% CI 2-sided [-46.0 to -22.8]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; Estimate Difference = -38.2, 95% CI 2-sided [-48.3 to -26.1]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; Estimate Difference = -49.3, 95% CI 2-sided [-57.7 to -39.4]

9. Secondary Outcome: Rate of Hypoglycemia With Blood Glucose <54 Milligram/Deciliter (mg/dL) [<3.0 Millimole/Liter (mmol/L)] or Severe Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with blood glucose <54mg/dL) (<3.0 mmol/L] or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. The rate of postbaseline hypoglycemia was estimated by negative binomial model: number of episodes = Pooled Country + Baseline Metformin Use (Yes, No) + Baseline HbA1c Group (<= 8.0%, >8.0%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline through Safety Follow-Up (Up to Week 44)
Population: All randomly assigned participants who took at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 116 | 119 | 120 | 120
Episodes/participant/365.25 days | 0.49 (0.141) | 0.66 (0.169) | 0.38 (0.099) | 0.51 (0.149)

10. Secondary Outcome: Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) of Tirzepatide
Description: AUC is a combined measure obtained from Week 7, 15, 23 and 39 and a single averaged measure of AUC was reported.
Time Frame: Week 7, 15, 23 and 39 post dose
Population: All randomized participants who received at least one dose and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 115 | 116 | 118
nanogram*hour per milliliter (ng*h/mL) | 79700 (24.5) | 164000 (26.7) | 246000 (26.4)

11. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target Value of <5.7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 40
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
Number analyzed (Participants) | 115 | 113 | 117 | 118
Percentage of Participants | 26.09 | 47.79 | 62.39 | 2.54
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.22, 95% CI 2-sided [3.93 to 38.00]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 32.36, 95% CI 2-sided [10.52 to 99.49]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 56.26, 95% CI 2-sided [18.27 to 173.26]

ADVERSE EVENTS:
Time Frame: Baseline, 17 Months
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/119 | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 9/116 | 13/119 | 9/120 | 10/120
Other Adverse Events (participants affected / at risk) | 52/116 | 60/119 | 67/120 | 58/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=116) | 10 mg Tirzepatide (N=119) | 15 mg Tirzepatide (N=120) | Placebo (N=120)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/55 (0) | 1/47 (1) | 0/55 (0) | 0/54 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic lesion excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=116) | 10 mg Tirzepatide (N=119) | 15 mg Tirzepatide (N=120) | Placebo (N=120)
Constipation (Gastrointestinal disorders) | 7 (7) | 8 (8) | 8 (9) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (22) | 15 (46) | 25 (44) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 10 (12) | 6 (6) | 2 (2)
Eructation (Gastrointestinal disorders) | 6 (11) | 4 (16) | 7 (11) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 6 (21) | 7 (12) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (26) | 21 (43) | 22 (44) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (12) | 9 (18) | 15 (26) | 3 (3)
Nasopharyngitis (Infections and infestations) | 18 (23) | 8 (11) | 15 (19) | 23 (27)
Lipase increased (Investigations) | 4 (4) | 2 (2) | 10 (12) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 15 (17) | 17 (21) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 16 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (4) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 6 (7) | 4 (6) | 7 (7)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 1 (1) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT04039503/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04039503/SAP_001.pdf